CLINICAL TRIAL: NCT01664247
Title: The Effect of Insulin Degludec in Combination With Liraglutide and Metformin in Subjects With Type 2 Diabetes Qualifying for Treatment Intensification
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3944; 2011-004665-32 (EudraCT Number); U1111-1124-6612 (Other: WHO)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg + Lira (Experimental)
  Interventions: Drug: insulin degludec; Drug: liraglutide
- Placebo + Lira (Experimental)
  Interventions: Drug: placebo; Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec — Administered s.c. (under the skin) once daily. Dose individually adjusted.
  Arms: IDeg + Lira
Drug: placebo — Administered s.c. (under the skin) once daily. Dose individually adjusted.
  Arms: Placebo + Lira
Drug: liraglutide — Administered s.c. (under the skin) once daily. Dose: 1.8 mg.

SUMMARY:
This trial is conducted in Africa, Asia, Europe and North America. The purpose of the trial is to investigate the effect of insulin degludec (IDeg) in combination with liraglutide (Lira) and metformin (at least 1500 mg daily or maximum tolerated dose) in subjects with type 2 diabetes qualifying for treatment intensification.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin naïve
* Ongoing treatment with metformin or metformin in combination with either sulphonylurea (SU), glinides, dipeptidyl peptidase-IV (DPP-IV) inhibitors or exenatide (only twice daily (BID))
* Glycosylated haemoglobin (HbA1c) (by central laboratory analysis): a. 7.5-10.0 % (both inclusive) for subjects on metformin monotherapy, b. 7.0-9.0 % (both inclusive) for subjects on metformin in combination with either SU, glinides, DPP-IV inhibitors or exenatide (only BID)

Exclusion Criteria:

* Treatment with glucose-lowering agent(s) other than stated in the inclusion criteria within 12 weeks
* Calcitonin equal to or above 50 pg/mL
* Stroke; heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty; all within 24 weeks
* Current or past (within the last 5 years) malignant neoplasms (except basal cell and squamous cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (120):
- United States (62):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (6):
  - Novo Nordisk Investigational Site, Delta, British Columbia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Québec
- France (11):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Mérignac
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Niort
  - Novo Nordisk Investigational Site, Pau
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Saint-denis de La Reunion
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (9):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Kirn
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Völklingen
- Israel (6):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (5):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Verona
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Novi Sad
- South Africa (4):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Ukraine (5):
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Lviv
  - Novo Nordisk Investigational Site, Ternopil
  - Novo Nordisk Investigational Site, Vinnitsa
- United Arab Emirates (4):
  - Novo Nordisk Investigational Site, Abu Dhabi
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Ras al-Khaimah
  - Novo Nordisk Investigational Site, Sharjah city
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Stevenage

REFERENCES:
- [Result] Aroda VR, Bailey TS, Cariou B, Kumar S, Leiter LA, Raskin P, Zacho J, Andersen TH, Philis-Tsimikas A. Effect of adding insulin degludec to treatment in patients with type 2 diabetes inadequately controlled with metformin and liraglutide: a double-blind randomized controlled trial (BEGIN: ADD TO GLP-1 Study). Diabetes Obes Metab. 2016 Jul;18(7):663-70. doi: 10.1111/dom.12661. Epub 2016 May 2. PMID 26990378
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 129 sites in 11 countries randomised subjects: Canada (7), France (10), Germany (8), Israel (6), Italy (7), Serbia (7), South Africa (6), Ukraine (4), United Arab Emirates (3), United Kingdom (6), and United States (65).
Groups:
- IDeg: Liraglutide treatment was initiated on 0.6 mg daily for one week and increased further after the second week in the run-in period. In the randomized period, Insulin degludec (IDeg, 100 U/mL, in a 3 mL prefilled pen PDS290) treatment was recommended to be initiated and administered subcutaneously (under the skin) once daily (OD) with 10 units. After that it was titrated once weekly. If one or more of the pre-breakfast plasma glucose values were below a certain range, the subjects were to reduce the insulin dose. Subjects continued on metformin (1500/day) treatment at the stable, pre-trial dose and maintained dosing frequency levels throughout the trial period.
- Placebo: Placebo treatment (3 mL prefilled pen) in combination with Liraglutide (Lira,1.8 mg/daily, 3 mL prefilled pen) once daily was given subcutaneously (under the skin) in the thigh, abdomen or upper arm (deltoid) at any time of the day according to the subject's choice for 26 weeks of treatment period. Subjects continued on metformin (1500/day) treatment at the stable, pre-trial dose and maintained dosing frequency levels throughout the trial period.
Period: Overall Study
Arm/Group | IDeg | Placebo
Started | 174 | 172
Exposed | 173 (1 subject was randomised in error and withdrew before exposure to the drug) | 170 (Two subjects were randomised in error and withdrew prior to exposure to drug)
Completed | 160 | 131
Not Completed | 14 | 41
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal Criteria | 1 | 4
Not completed — Unclassified | 5 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg | Placebo | Total
Number analyzed (Participants) | 174 | 172 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.0) | 57.3 (9.4) | 57.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 68 | 144
  Male | 98 | 104 | 202
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.5 (0.6) | 7.6 (0.6) | 7.6 (0.6)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.7 (2.1) | 9.1 (2.2) | 8.9 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) (%)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 174 | 172
percentage of glycosylated haemoglobin | -0.99 (0.08) | -0.07 (0.08)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 6 subjects FPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 172 | 168
mmol/L | -2.60 (2.91) | -0.28 (2.44)

3. Secondary Outcome: Number of Responders for HbA1c (Below 7.0 %)
Description: Number of responders for HbA1c below 7.0%, after 26 weeks of randomised treatment.
Time Frame: After 26 weeks of randomised treatment.
Population: The FAS included all randomised subjects and missing data was imputed using LOCF.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 174 | 172
percentage (%) of subjects | 77.6 | 35.5

4. Secondary Outcome: Change From Baseline in Mean Pre-breakfast Measurements Used for Titration
Description: Change from baseline after 26 weeks of treatment in the average of the pre-breakfast self measured plasma glucose (SMPG) measured on the day of the contact and the two days immediately prior to the contact. The least squares means presented are the estimated values after 26 weeks of treatment and the statistical analysis presents the treatment difference of the change from baseline values as the model is adjusted for baseline.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 8 subjects the baseline values were missing
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 171 | 167
mmol/L | 5.88 (0.14) | 8.23 (0.15)
Statistical Analysis 1: Comparison: IDeg vs Placebo; The pre-breakfast measures of SMPG values after 26 weeks of treatment were analysed an ANOVA method with treatment, region and sex as fixed effects, and age and baseline response as covariates; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-2.67 to -2.01] — The treatment contrast estimated was IDeg - Placebo

5. Secondary Outcome: Change From Baseline in 8-point Profile
Description: The change from baseline in the 8-point SMPG profile after 26 weeks of randomised treatment. The least squares means presented are the estimated values after 26 weeks of treatment and the statistical analysis presents the treatment difference of the change from baseline values as the model is adjusted for baseline.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. The subjects not analysed were 12, 45, 46, 44, 44, 54, 56 and 21 subjects for before breakfast, 90 mins after breakfast, before lunch, 90 mins after start of lunch, before main evening meal, 90 mins after main evening meal, before bedtime and before breakfast the following day time points respectively.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 172 | 169
mmol/L
  Before breakfast, N=170, 164 | 5.85 (0.15) | 8.54 (0.16)
  90 min after breakfast, N=153, 148 | 7.65 (0.24) | 9.75 (0.25)
  Before lunch, N=151,149 | 6.33 (0.18) | 8.34 (0.19)
  90 min after lunch, N=152,150 | 7.73 (0.21) | 9.67 (0.21)
  Before evening meal, N=154,148 | 6.77 (0.20) | 9.51 (0.21)
  90 mins after evening meal, N=147,145 | 7.93 (0.21) | 9.65 (0.22)
  Before bedtime, N=148, 142 | 7.21 (0.20) | 8.95 (0.21)
  Before breakfast the next day, N=164,161 | 6.05 (0.17) | 8.55 (0.18)
Statistical Analysis 1: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point before breakfast; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-3.04 to -2.34] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 2: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point 90 mins after breakfast; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-2.71 to -1.48] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 3: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point before lunch; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.01, 95% CI 2-sided [-2.47 to -1.56] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 4: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point 90 mins after start of lunch; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Median Difference (Final Values) = -1.93, 95% CI 2-sided [-2.46 to -1.40] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 5: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point main evening meal; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-2.25 to -1.23] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 6: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point 90 mins after main evening meal; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.26 to -1.18] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 7: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point before bedtime; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-2.27 to -1.23] — The treatment contrast estimated was IDeg - Placebo
Statistical Analysis 8: Comparison: IDeg vs Placebo; The 8-point profile (SMPG) values after 26 weeks of treatment were analysed jointly using a linear mixed model with an un-structured residual covariance structure and with treatment, time-point and an interaction between treatment and time-point, region and sex as fixed effects, and age and baseline response per time-point as covariates. Missing data was imputed using LOCF. The treatment contrast estimated was IDeg - Placebo for the time point before breakfast the following day; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-2.91 to -2.09] — The treatment contrast estimated was IDeg - Placebo

6. Secondary Outcome: Change From Baseline in Mean of the 8-point Profile
Description: Change from baseline in mean of the 8-point profile after 26 weeks of randomised treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data is imputed using LOCF. Mean values were missing for 11 subjects.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 169 | 166
mmol/L | -2.3 (1.8) | -0.5 (1.7)

7. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Number of confirmed hypoglycaemic episodes from week 0 to 26 weeks of randomised treatment. A hypoglycaemic episode was defined as treatment emergent if the onset of the episode occurred after the first administration of investigational medicinal product and no later than 7 days after the last day on trial product. Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia or minor hypoglycaemic episodes.
Time Frame: Weeks 0 - 26
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 173 | 170
events | 47 | 9

8. Secondary Outcome: Number of Adverse Events
Description: Number of treatment emergent AEs (TEAEs) from week 0 to week 26 of the randomised treatment. A TEAE was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Weeks 0 - 26
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 173 | 170
events | 285 | 252

9. Secondary Outcome: Change From Baseline in Patient Reported Health-related Quality of Life Using the Short-Form 36 Health Survey Version 2 (SF-36®v2)
Description: Change in subject's quality of life was evaluated using the Short-Form 36 Health Survey version 2 (SF-36®v2). Evaluations were performed at baseline and at the last treatment visit (week 26). SF-36 was assessed on a scale range of 0.65 to 80.73 for physical health and -8.81 to 81.65 for mental health respectively, where higher scores indicated a better quality of life. 0-100 scores from the SF-36 were converted to a norm-based score using a T-score transformation in order to obtain a direct interpretation in relation to the distribution of the scores in the 1998 U.S. general population.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 3 subjects PRO scores were missing at the baseline and did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | IDeg | Placebo
Number analyzed (Participants) | 174 | 169
T-scores
  Physical health | 0.5 (6.3) | 0.0 (6.2)
  Mental health | 0.6 (8.1) | -0.7 (8.8)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up. Adverse event with an onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/173 | 9/170
Other Adverse Events (participants affected / at risk) | 33/173 | 32/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=173) | Placebo (N=170)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lentigo maligna stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=173) | Placebo (N=170)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 13 (17)
Nasopharyngitis (Infections and infestations) | 14 (15) | 11 (12)
Lipase increased (Investigations) | 10 (11) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.